CLINICAL TRIAL: NCT04170764
Title: Clinical Utility of Postoperative Hemoglobin Testing Following Vaginal Hysterectomy and Reconstruction for Symptomatic Pelvic Organ Prolapse
Brief Title: Clinical Utility of Postoperative Hemoglobin Testing
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 19-111
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-10

CONDITIONS: Anaemia Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate how many patients have hemoglobin less than 10 g/dL at post-operative day 1

DETAILED DESCRIPTION:
Obtaining a complete blood count (CBC) on post-operative day 1 to assess postoperative hemoglobin levels is routine practice at Cincinnati Urogynecology Associates, TriHealth Inc. after pelvic reconstructive surgery.

There is minimal data supporting this practice. Multiple studies throughout the gynecology literature suggest that this is not a necessary or cost effective strategy to assess for postoperative anemia. Most patients who require blood transfusion or reoperation for bleeding will show clinical signs of anemia.

The investigators aim to determine if checking a routine CBC results in clinically relevant changes to patient care in women undergoing pelvic reconstructive surgery with vaginal hysterectomy for treatment of pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Total vaginal hysterectomy with or without bilateral salpingectomy/oophorectomy (CPT 58260, 58262, 58263, 58270, 58290, 58291, 58292, 58294)
* At least one of the following vaginal native tissue prolapse repairs

  * Apical repair with uterosacral ligament suspension (CPT 57283)
  * Apical repair with sacrospinous ligament fixation (CPT 57282)
  * Anterior repair (CPT 57240, 57260, 57284, 57285, 57250)
  * Posterior repair (CPT 45560, 56800, 56810, 57200, 57210, 57250)
* Surgery by one of four fellowship trained urogynecologists at TriHealth

Exclusion Criteria:

* Concomitant surgical procedure by a second surgeon
* Malignancy identified at the time of surgery or active malignancy
* Cases converted to open hysterectomy or prolapse repairs
* Prolapse repair completed robotically
* Prolapse repair completed with mesh
* Known coagulopathy
* Patient on long term preoperative anticoagulant medication (Arixtra, Coumadin, Eliquis, Heparin, Lovenox, Pradaxa, Savaysa, Xarelto)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent a total vaginal hysterectomy with concurrent vaginal native tissue prolapse repairs performed by one of four fellowship trained urogynecologists at TriHealth between 10/1/2014 and 10/1/2019. The patients will be identified by CPT codes in the EPIC electronic medical record.
Sampling Method: Non-Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Aldrich ER, Pauls RN. Clinical Benefit of Routine Postoperative Hemoglobin Testing After Vaginal Hysterectomy and Reconstruction for Symptomatic Pelvic Organ Prolapse. Female Pelvic Med Reconstr Surg. 2022 Jan 1;28(1):40-44. doi: 10.1097/SPV.0000000000001056. PMID 33787565

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaginal Hysterectomy With Reconstruction: All patients who underwent a total vaginal hysterectomy with concurrent vaginal native tissue prolapse repairs performed by one of four fellowship trained urogynecologists at TriHealth between 10/1/2014 and 10/1/2019.
  The patients will be identified by CPT codes in the EPIC electronic medical record.
Period: Overall Study
Arm/Group | Vaginal Hysterectomy With Reconstruction
Started | 664
Completed | 571
Not Completed | 93

BASELINE CHARACTERISTICS:
Arm/Group | Vaginal Hysterectomy With Reconstruction
Number analyzed (Participants) | 573
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.22 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 573
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 533
  African American | 23
  Hispanic | 8
  Asian | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 573

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With POD1 Hemoglobin Less Than 10 g/dL
Time Frame: Postop Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Hysterectomy With Reconstruction
Number analyzed (Participants) | 571
Participants | 97

ADVERSE EVENTS:
Time Frame: POD 1
Arm/Group | Vaginal Hysterectomy With Reconstruction
All-Cause Mortality (participants affected / at risk) | 0/571
Serious Adverse Events (participants affected / at risk) | 0/571
Other Adverse Events (participants affected / at risk) | 0/571

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT04170764/Prot_SAP_000.pdf